CLINICAL TRIAL: NCT03506542
Title: Phacotrabeculectomy With Collagen Matrix Implant (Ologen®) Versus Mitomycin C Augmented Phacotrabeculectomy: Clinical Results of a Prospective Randomized Trial
Brief Title: Phacotrabeculectomy With Collagen Matrix Implant (Ologen®) Versus Mitomycin C
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of Lublin (Other)
Collaborators: Aeon Astron Europe B.V. (Industry)
Responsible Party: Principal Investigator, Aleksandra Wlaz, PhD, ophthalmologist in Department of Diagnostics and Microsurgery of Glaucoma, Medical University of Lublin
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: not required
Record Dates: First submitted 2018-04-14; First posted 2018-04-24 (Actual); Last update posted 2018-04-25 (Actual); Status verified 2018-04

CONDITIONS: Glaucoma; Cataract; Wound Heal
MeSH Terms: conditions — Glaucoma; Cataract | interventions — Surgical Procedures, Operative; Mitomycin

STUDY DESIGN:
Intervention Model Description: Patients are randomized and have phacotrabeculectomy augmented with either OLO (Ologen) or MMC (Mitomycin C).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Ologen (OLO) (Experimental): Ologen implant (model 830601) placed over scleral flap during phacotrabeculectomy
  Interventions: Device: Ologen; Procedure: Phacotrabeculectomy
- Mitomycin C (MMC) (Active Comparator): Mitomycin C (MMC) 0.3 mg/ml for 3 minutes under the scleral flap during phacotrabeculectomy (standard procedure)
  Interventions: Procedure: Phacotrabeculectomy; Drug: Mitomycin C

INTERVENTIONS:
Device: Ologen — Ologen implant placed over scleral flap during the surgery to avoid usage of Mitomycin C
  Other Names: OLO
  Arms: Ologen (OLO)
Procedure: Phacotrabeculectomy — Trabeculectomy with cataract extraction
  Other Names: surgery
Drug: Mitomycin C — Mitomycin C 0.3 mg/ml for 3 minutes during the surgery (standard procedure)
  Other Names: MMC
  Arms: Mitomycin C (MMC)

SUMMARY:
1. Study objective: To assess the efficacy and safety of collagen matrix implant (Ologen®; OLO) in phacotrabeculectomy and to compare with mitomycin C (MMC) augmented phacotrabeculectomy.
2. Study Design: The study is designed as a prospective randomized trial. Patient who meet the inclusion/exclusion criteria and sign the informed consent form will be included for this study.
3. Follow-Up: This investigation is including 7 post-operative visits and follow-up within 12 months from the date of surgery. Patients should be seen at postoperative days 1, 7, 30, 90, 180, 270 and 360.

DETAILED DESCRIPTION:
* Prospective randomized comparative study
* Patients with cataract and:

primary open angle glaucoma (POAG) pseudoexfoliation (PEX) glaucoma (PEXG)

* Phacotrabeculectomy augmented with OLO or MMC
* Follow-up - 12 months

ELIGIBILITY:
Inclusion Criteria:

* Cataract
* Primary open angle glaucoma or pseudoexfoliation glaucoma with progression of visual field loss and/or uncontrolled intraocular pressure levels with medication

Exclusion Criteria:

* Difficulty in reading or speaking Polish
* Previous ocular surgery
* Pregnant and breastfeeding women
* Angle closure glaucoma
* Secondary glaucoma except pseudoexfoliation glaucoma
* Ocular diseases with excessive scarring
* Allergy to collagen or Mitomycin C

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2014-06-02 (Actual); Primary Completion 2016-03-01 (Actual); Study Completion 2017-03-30 (Actual)

PRIMARY OUTCOMES:
Mean intraocular pressure (IOP) after the surgery | 12 months
  Decrease in IOP before and after the surgery

SECONDARY OUTCOMES:
Mean best corrected visual acuity (BCVA) (LogMAR) | 12 months
  Increase in best corrected visual acuity (BCVA) (LogMAR) before and after the surgery
Evaluation of the filtering bleb in MBGS (Moorfields Bleb Grading System) | 12 months
  To compare filtrating blebs in two arms of the study
Mean number of antiglaucoma medications | 12 months
  To compare the number of antiglaucoma medications in two arms of the study

CONTACTS AND LOCATIONS:
Overall Officials: Tomasz Żarnowski, MD PhD Prof, Study Chair — Ophthalmology Clinic, Medical University in Lublin, Poland